CLINICAL TRIAL: NCT06994403
Title: Evaluation of the Glycemic Response to a Pasta Enriched With Carob Flour: a Study Conducted in Healthy Subjects and a Study Conducted in Subjects With Type 1 Diabetes Mellitus
Brief Title: Glycemic Response to Carbob-Enriched Pasta in Healthy and With Type 1 Diabetes People
Acronym: GR-CEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Lutgarda Bozzetto, Professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 32/2023
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Glycemic and Insulinemic Response; Type 1 Diabetes (T1D)
Keywords: Ceratonia siliqua; Glycemic Index; Type 1 Diabetes; Functional Foods; Postprandial Glycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — locust bean gum

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carob-Enriched Durum Wheat Pasta (Experimental): Participants will consume 68 g of carob-enriched durum wheat pasta (231 kcal) containing 50 g of available carbohydrates, served with 55 g of tomato sauce prepared with 2.5 g of extra virgin olive oil.
  Interventions: Dietary Supplement: Durum wheat pasta enriched with carob flour; Dietary Supplement: Standard durum wheat pasta; Dietary Supplement: White bread reference meal
- Durum Wheat Pasta (Sham Comparator): Participants will consume 63 g of traditional durum wheat pasta (221 kcal) containing 50 g of available carbohydrates, served with 55 g of tomato sauce prepared with 2.5 g of extra virgin olive oil.
  Interventions: Dietary Supplement: Durum wheat pasta enriched with carob flour; Dietary Supplement: Standard durum wheat pasta; Dietary Supplement: White bread reference meal
- White Bread (Reference Food) (Active Comparator): Participants will consume 84 g of white bread (225 kcal) containing 50 g of available carbohydrates, served with 55 g of tomato sauce prepared with 2.5 g of extra virgin olive oil.
  Interventions: Dietary Supplement: Durum wheat pasta enriched with carob flour; Dietary Supplement: Standard durum wheat pasta; Dietary Supplement: White bread reference meal

INTERVENTIONS:
Dietary Supplement: Durum wheat pasta enriched with carob flour — Participants will consume 68 g of durum wheat pasta enriched with carob flour (231 kcal), providing 50 g of available carbohydrates. The pasta will be served with 55 g of tomato sauce prepared with 2.5 g of extra virgin olive oil.
Dietary Supplement: Standard durum wheat pasta — Participants will consume 63 g of standard durum wheat pasta (221 kcal), providing 50 g of available carbohydrates. The pasta will be served with 55 g of tomato sauce prepared with 2.5 g of extra virgin olive oil.
Dietary Supplement: White bread reference meal — Participants will consume 84 g of white bread (225 kcal), providing 50 g of available carbohydrates. The bread will be served with 55 g of tomato sauce prepared with 2.5 g of extra virgin olive oil.

SUMMARY:
Carob (Ceratonia siliqua) is a fruit traditionally used in various Mediterranean countries for the preparation of sweets and beverages. Its pulp, once the seeds are removed, is milled into carob flour, a nutrient-rich food containing fiber, carbohydrates, proteins, and essential minerals such as potassium, magnesium, sodium, phosphorus, and calcium. Carob flour is also naturally sweet and can serve as a cocoa powder substitute in desserts. Furthermore, it is a source of polyphenols with known antioxidant properties.

Clinical evidence suggests that consumption of foods rich in refined carbohydrates is associated with elevated postprandial blood glucose levels, which are recognized as an independent cardiovascular risk factor. The glycemic index (GI) is a useful parameter to assess the impact of carbohydrate-containing foods on postprandial glycemic response. Based on carbohydrate quality, foods are classified as having high, medium, or low GI. Consumption of high-GI foods leads to a stronger glycemic response and has been linked to increased risk of chronic conditions such as type 2 diabetes, obesity, and cardiovascular disease.

Given its bromatological profile, carob flour may have the potential to modulate postprandial glycemic responses. However, studies evaluating the GI of carob-based products have shown inconsistent findings. In one randomized trial involving 10 healthy adults, a carob-based snack demonstrated a lower GI (40) compared to a chocolate cookie with an equivalent carbohydrate content (GI 78), using glucose as the reference. The same study found that consuming the carob snack before a meal led to a reduced postprandial glycemic response, decreased hunger, and lower caloric intake at an ad libitum meal. Another study on 7 healthy individuals reported a GI of 39 for carob flour bars containing 26 g of available carbohydrates. Conversely, a study involving 20 healthy participants found that consuming 5 or 10 g of carob pulp with 200 mL of water and 50 g glucose increased postprandial glycemic and insulinemic responses compared to water and glucose alone. This effect was not observed with a 20 g dose of carob pulp.

Among carbohydrate-rich foods, pasta represents a key component of the Italian diet and, due to its physical structure, generally has a low-to-moderate GI. Compared to other wheat-based foods like bread, pasta tends to produce a lower postprandial glycemic response when carbohydrate content is matched. However, the impact of adding carob flour to durum wheat semolina in pasta production on postprandial glycemia remains unexplored.

The current research project consists of two studies. The first study aims to determine the glycemic index of carob-enriched durum wheat pasta in healthy adult volunteers, using white bread as the reference food. The second study investigates the postprandial glycemic response to the same carob-enriched pasta in individuals with type 1 diabetes, comparing it to traditional durum wheat pasta. These studies are designed to contribute to the understanding of carob flour's role in glycemic control, with potential implications for dietary management in both healthy individuals and patients with diabetes.

DETAILED DESCRIPTION:
Study 1:

This randomized, controlled, crossover trial aims to determine the glycemic index (GI) of a durum wheat pasta enriched with carob flour in healthy adult males. Over a period of three months, participants will consume test meals on separate days under controlled conditions. The glycemic response will be compared to that elicited by white bread, which serves as the reference food. This study is conducted in an outpatient setting and will contribute to the evaluation of the metabolic impact of carob-enriched pasta on postprandial glycemia.

Study 2:

This controlled, crossover study is designed to assess the postprandial glycemic response to carob flour-enriched pasta in individuals with type 1 diabetes using continuous glucose monitoring (CGM). Conducted over a 12-month period, the study involves alternating consumption of carob-enriched and standard durum wheat pasta. Participants will follow their usual dietary habits while maintaining consistent meal composition and daily routines during the test days. The study aims to explore the potential of carob-enriched pasta to modulate postprandial glycemia in a population with impaired glucose regulation.

ELIGIBILITY:
Inclusion Criteria:

Study 1

* Healthy male volunteers
* Age between 18 and 50 years
* Body Mass Index (BMI) between 18 and 29 kg/m²

Study 2

* Male and female individuals
* Age ≥ 18 years
* Confirmed diagnosis of type 1 diabetes mellitus
* Use of a continuous glucose monitoring (CGM) system

Exclusion Criteria:

Study 1

* Diagnosis of diabetes mellitus
* Presence of any chronic-degenerative disease
* Any acute or chronic medical condition that could seriously compromise overall health
* Diagnosis of celiac disease

Study 2

* Presence of serious chronic illnesses (e.g., coronary heart disease, renal failure, liver diseases, endocrine disorders)
* Gastrointestinal disorders
* Pregnancy or breastfeeding
* Alcohol or drug dependence

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Glycemic Index of Carob-Enriched Durum Wheat Pasta | Within 2 hours after consumption of the test meal on three separate test days (each separated by at least 2 days).
  The primary outcome is the determination of the glycemic index (GI) of a carob-enriched durum wheat pasta compared to white bread, used as the reference food. The glycemic response will be assessed through blood glucose concentrations measured at fasting and at 15, 30, 60, 90, and 120 minutes after consumption.

OTHER OUTCOMES:
Postprandial Glycemic Response (iAUC) to Carob-Enriched Pasta in Type 1 Diabetes | 6 hours post-meal on 6 different test days over a 2-week period.
  The outcome is the incremental area under the curve (iAUC) of postprandial blood glucose levels measured by continuous glucose monitoring (CGM) after consumption of carob-enriched durum wheat pasta, compared to standard durum wheat pasta. Glucose data will be analyzed in the 30 minutes before and 6 hours after meal intake.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppina Costabile, Study Chair — Federico II University
Locations (1):
- Federico II University, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol